CLINICAL TRIAL: NCT07230886
Title: Prospective Reduction Of Transplant Complications Through Enhanced Preservation Therapy to Prevent Primary Graft Dysfunction
Acronym: PROTECT-PGD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: CareDx (Industry); Montreal Heart Institute (Other); London Health Sciences Centre (Other); Ottawa Heart Institute Research Corporation (Other); Traferox Technology Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 25-5039
Record Dates: First submitted 2025-08-12; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-08

CONDITIONS: Primary Graft Dysfunction
Keywords: Primary Graft Dysfunction; Transplant; Traferox; Preservation Therapy; X Port Preservation System
MeSH Terms: conditions — Primary Graft Dysfunction

STUDY DESIGN:
Intervention Model Description: multicentre, feasibility, randomized, blinded, controlled pilot trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participant and all study personnel will be blinded to the treatment arm the participant is randomized to - with exception to the unblinded research assistant that will be performing the randomization and allocation process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xo Port Organ Preservation System (Experimental): Traferox Transport System containing eutectic gel-packs used for controlled hypothermic storage
  Interventions: Device: Xo Port Organ Preservation System
- Static Ice Storage (Active Comparator): Traferox Transport System containing ice-packs as used for conventional cold static storage
  Interventions: Device: Standard of Care - Ice packs

INTERVENTIONS:
Device: Xo Port Organ Preservation System — It is a disposable temperature-controlled hypothermic transportation system that maintains the donated heart temperature between 8 and 12°C. It consists of an insulated chamber; eutectic gel packs containing a specialized phase change material (composition under manufacturer's patent) preconditioned before use (by freezing in a 4°C temperature-regulated refrigerator for 48 hours), which maintain temperature between 8 and 12°C through passive cooling; a removable insert, a cradle to hold the organ bag, an internal temperature probe; a logger for continuous monitoring and maintenance of temperature over an extended period of time, an internal venting system that allows air circulation to ensure homogenous temperature for a validated maximal time of 24 hours; and casters and a telescopic handle to facilitate transport.
  Other Names: Traferox Transport System
  Arms: Xo Port Organ Preservation System
Device: Standard of Care - Ice packs — Cold static donor heart preservation is currently the mainstay of organ transportation after procurement. The donor heart is placed in the Traferox Transport system with ice-packs.
  Arms: Static Ice Storage

SUMMARY:
The goal of this clinical trial is to test the feasibility of the study protocol comparing a novel temperature control system - Xo Port Organ Preservation System - to static ice for heat preservation for Heart Transplant. The main questions of the study are as follows:

Does the Incidence of severe PGD change within the first 24 hours of heart transplant in patients randomized to the Xo Port Organ Preservation System?

Was there a change in composite efficacy endpoints in participants randomized to the Xo Port Organ Preservation System compared to static ice storage?

Were the feasibility outcomes achieved?

Were there any protocol deviations?

Participants will:

Be randomized to either the Xo Port Organ Preservation System or static ice storage.

Complete a questionnaire at the time of screening, day 0, 7, and 90 days post transplant.

Have blood drawn - with their standard of care blood draws - after their transplant, the day after, and 7 days post transplant.

DETAILED DESCRIPTION:
The PROTECT-PGD Pilot trial is a 2.5 year, 50-patient, multi-centre, feasibility, randomized, blinded, controlled pilot trial assessing feasibility of a full-scale blinded randomized controlled trial to determine whether use of the Xo Port Organ Preservation System (Traferox Technologies Inc.), a novel temperature controlled system that maintains donor heart temperature between 8 and 12°C reduces the risk of severe PGD in patients post HT. If feasibility is demonstrated, pilot trial participants will be included in the full-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Recipient: Adult (>17 years old)
* Donor: Donation after brain death acceptable for transplant as determined by a procuring physician unaware of randomization sequence at the time of acceptance

Exclusion Criteria:

* Recipient: Multi-organ transplant recipients; Participating in an interventional study.
* Donor: Donation after cardiac death; Use of organ care system

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Primary Study Feasibility | 2.5 years
  Determined by the mean number of participants recruited per month calculated on recruitment over 24 months.
Composite efficacy outcome of full-scare trial 1 | 2.5 years
  90-day mortality
Composite efficacy outcome of full-scare trial 2 | 2.5 years
  severe PGD (defined through the ISHLT consensus definition need for MCS will be adjudicated in a blinded fashion with LVEF<40% and CI<2.0 on high dose inotropes
Composite efficacy outcome of full-scare trial 3 | 2.5 years
  duration of mechanical ventilation
Composite efficacy outcome of full-scare trial 4 | 2.5 years
  ICU length of stay (LOS)
Composite efficacy outcome of full-scare trial 5 | 2.5 years
  index transplant LOS
Composite efficacy outcome of full-scare trial 6 | 2.5 years
  Moderate to severe rejection based on ISHLT criteria at 90 days
Composite efficacy outcome of full-scare trial 7 | 2.5 years
  change in EQ-5D-5L utility index score from baseline to 90 days with a clinically meaningful change defined as >0.05
Composite efficacy outcome of full-scare trial 8 | 2.5 years
  cfDNA count measured over POD0, POD1, and POD7

CONTACTS AND LOCATIONS:
Overall Officials: Yasbanoo Moayedi, MD, Principal Investigator — University Health Network, Toronto